CLINICAL TRIAL: NCT05126563
Title: A Randomized, Double-blinded, Single-center, Phase 2 Efficacy, and Safety Study of Allogeneic HB-adMSCs for the Treatment of Patients With Chronic Post-COVID-19 Syndrome.
Brief Title: Randomized Double-Blind Phase 2 Study of Allogeneic HB-adMSCs for the Treatment of Chronic Post-COVID-19 Syndrome
Acronym: HBPCOVID02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HBPCOVID02
Record Dates: First submitted 2021-11-12; First posted 2021-11-19 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Post COVID-19 Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Double-Blind
Who Masked: Participant, Care Provider, Investigator
Masking Description: Amber bags will be used to 'blind' the participant and investigator to which group the subject belongs in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): HB-ad MSC's allogeneic
  Interventions: Biological: HB-adMSCs (allogeneic)
- Placebo (Placebo Comparator): Sterile Normal Saline
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: HB-adMSCs (allogeneic) — HB-adMSCs allogenic
  Other Names: Hope Biosciences adipose derived mesenchymal stem cells
  Arms: Treatment
Other: Placebo — Placebo comarator
  Other Names: Sterile Normal Saline
  Arms: Placebo

SUMMARY:
This study will enroll up to 80 subjects with Chronic Post COVID-19 Syndrome. Subjects will receive four intravenous injections of either allogeneic HB-adMSC's or a placebo over 10 weeks with two follow-up visits and an end of study visit at week 26.

DETAILED DESCRIPTION:
Active Product: HB- adMSCs (Hope Biosciences adipose-derived mesenchymal stem cells - allogeneic) Dose: 200 million Route: Intravenous Regimen: Weeks 0, 2, 6, and 10. Placebo: Saline Solution 0.9% Dose: N/A Route: Intravenous Regimen: Weeks 0, 2, 6, and 10.Duration of administration 1 hour Laboratory Samples. Screening, Week 0, 6, and 26. Visits by Weeks Screening Week 0 - Infusion 1 Week 2 - Infusion 2 Week 6 - Infusion 3 Week 10 - Infusion 4 Week 14 - Follow Up 1 Week 20 - Follow Up 2 Week 26 - End of Study

ELIGIBILITY:
Inclusion Criteria:

A study participant will be eligible for inclusion in this study only if all the following criteria apply:

1 Male and female participants 18 - 70 years of age.

2. Participants in the study have proof of Post COVID-19 Syndrome in their medical records.

3. Study participants must have been diagnosed with Chronic post-COVID-19 syndrome for at least twelve weeks before enrollment in the clinical trial.

4. The study participant is experiencing one or more neurological symptoms for at least 12 weeks, either continually or intermittently, with relapses not experienced pre-illness that interferes with regular daily activities. Symptoms must be new symptoms or dramatic worsening of preexisting symptoms, i.e., the subject didn't have symptoms and had not sought medical treatment for the symptoms before COVID-19, or the symptoms are dramatically worse (in severity and frequency). At least one symptom must have a severity of "5cm" on the neurological symptom VAS at screening. See the list of symptoms below:

* Extreme fatigue: Feeling overtired with low energy and a strong desire to sleep.
* Brain Fog: A diminished mental capacity marked by the inability to concentrate, think or reason clearly interferes with daily activities.
* Headache: Sharp or dull reoccurring or intermittent that were not present pre-illness.
* Sleep Issues: Any sleep disturbances in sleep quality that makes sleep seem inadequate or unrefreshing like insomnia or hypersomnia.
* Loss of Taste/Smell: A diminished sense of taste or smell.

  5. Study participants should be able to read, understand, and provide written consent.

  6. Female study participants should not be pregnant or plan to become pregnant during study participation and six months after the last investigational product administration.

  7. If their sexual partners can become pregnant, male participants should use a method of contraception during study participation and for six months after the last administration of the experimental drug. *

  8. The study participant is able and willing to comply with the requirements of this clinical trial.

Exclusion Criteria:

A study participant will not be eligible for inclusion in this clinical trial if any of the following criteria apply:

1. The subject is unable to provide informed consent or to comply with study requirements.
2. A study participant has currently been diagnosed with active COVID-19 disease, defined as ongoing symptoms related to acute infection (such as fever or chills, cough, shortness of breath, or difficulty breathing, among other symptoms), and evidence of a positive RT-PCR SARS- CoV-2.
3. The subject is unwilling to agree to the use of acceptable methods of contraception * throughout the study and for six months after the last dose of the investigational product.
4. Pregnancy, lactation. Women of childbearing age who are not pregnant but do not take adequate contraceptive measures. *
5. The study participant has a history of addiction or dependency, or he or she is currently abusing or using substances.
6. Study participant has any active malignancy, including but not limited to evidence of cutaneous basal, squamous cell carcinoma, or melanoma.
7. The study participant has one or more significant concurrent medical conditions (verified by medical records), including the following:

   * Diabetes Mellitus (DM) Poorly controlled diabetes mellitus (PCDM), defined as a history of deficient standard of care treatment or pre-prandial glucose >130mg/dl during screening visit or post-prandial glucose >200mg/dl.
   * Chronic kidney disease (CKD): Medical History of Chronic kidney disease (CKD) diagnosis or screening results of eGFR < 59mL/min/1.73m2. Subjects with any form of kidney dialysis will be excluded from participation in this clinical trial.
   * Heart Failure Presence of New York Heart Association (NYHA) Class III/IV heart failure during the screening visit.
   * Myocardial Infarction: Medical history of myocardial infarction in any of the different types, such as ST-elevation myocardial infarction (STEMI) or non-ST-elevated myocardial infarction (NSTEMI), coronary spasm, or unstable angina.
   * High Blood Pressure: Medical history of uncontrolled high blood pressure is defined as a deficient standard of care treatment or blood pressure > 140/90 mm/Hg during the screening visit in a patient taking anti-hypertensive treatment. At screening visit, all patients must have a blood pressure <140/90 mmHg.
   * Other diseases: Medical history of inherited thrombophilias, cancer of the lung, brain, lymphatic, gynecologic system (ovary or uterus), or gastrointestinal tract (like pancreas or stomach).
   * Other conditions: Lower extremity paralysis due to spinal cord injury, fracture of the pelvis, hips or femur or recent major general surgery (within 12 months before the Screening).
8. Study participant has received any stem cell treatment within 12 months before the first dose of the investigational product other than stem cells produced by Hope Biosciences.
9. The study participant has received an experimental drug within 12 months before the first dose of the investigational product. (Except for COVID-19 vaccinations)
10. Study participant has a laboratory abnormality during screening, including the following:

    * White blood cell count WBC < 3.0 K/UL and > 12.0 K/UL
    * Platelet count < 80 K/UL and or > 450 K/UL
    * Absolute neutrophil count < 1.50 K/UL and or > 7.50 K/UL
    * Alanine aminotransferase (ALT) of > 75 U/L
    * Aspartate aminotransferase (AST) of > 75 U/L
    * Hemoglobin (Hgb) <11 G/DL or >18 G/DL
    * Hematocrit (HCT) <33% or >54 %
    * Mean corpuscular volume (MCV) < 75 FL or >100 FL
    * Mean corpuscular hemoglobin (MCH) <23 PG or >36 PG
    * Mean corpuscular hemoglobin concentration (MCHC) <30 G/DL or > 37gG/DL
    * Red cell distribution width (RDW) < 10% or >14%
    * Abnormal laboratory results considered clinically significant by the principal investigator will exclude patients from participation in this investigation.
11. The study participant has any known ongoing infection, including TB, CMV, EBV, HSV, VZV, hepatitis virus, toxoplasmosis, HIV, syphilis infections, hepatitis B surface antigen-positive, or hepatitis C PCR positivity.
12. The study participant is unlikely to complete the study or adhere to the study procedures.
13. The study participant has a previously diagnosed psychiatric condition that may affect self-assessments in the investigator's opinion.
14. Study participants with any systemic infection requiring treatment with antibiotics, antivirals, or antifungals within 30 days before the first dose of the investigational product.
15. Male study participants expect to donate sperm during the trial or within six months after the last dose. Female patients intend to donate eggs or have IVF treatment during the trial or within six months after the last dose.
16. Study participants who the Investigator determines to be unsuitable for study enrollment for other reasons, such as, but not limited to deep vein thrombosis (DVT), pulmonary embolus, those who have a prothrombotic condition, or who require persistent oxygen supplementation.
17. The subject has recently been diagnosed with an unstable Chronic obstructive pulmonary disease (COPD) as defined by patients who experience frequent or severe exacerbations and a faster decline in pulmonary function.
18. Subjects who have fatigue due to chronic kidney disease, iron deficiency anemia, B12 deficiency and other anemias will be excluded.
19. Any participant who has suicidal ideation at the screening visit will be excluded from this clinical trial.
20. Subjects with the following diseases must be excluded from participation in the trial.

    * chronic liver disease
    * pneumonia
    * history of chronic fatigue syndrome
    * subjects with fatigue symptoms due to fibromyalgia, arthritic disorders, inflammatory and rheumatological disorders
    * respiratory failure
    * emphysema
    * uncontrolled asthma
    * any subject requiring supplemental oxygen for any cause.

      * Acceptable reversible and permanent methods of birth control include:

1. True sexual abstinence (abstaining from sexual activity during the entire period of risk).

2. Surgery (occlusion bilateral tubal ligation, vasectomized partner). 3. Hormonal contraceptives associated with ovulation inhibition (oral, injectable, implantable patch, or intravaginal). 4. Intrauterine device (IUD), or intrauterine hormone-releasing system (IUS). 5. Condoms.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thanh Cheng, MD, Principal Investigator — Hope Biosciences Research Foundation
Locations (1):
- Hope Biosciences Research Foundation, Sugar Land, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- HB-adMSCs: HB-adMSCs (allogeneic): HB-adMSCs allogenic
Period: Overall Study
Arm/Group | HB-adMSCs | Placebo
Started | 39 | 40
Completed | 34 | 30
Not Completed | 5 | 10

BASELINE CHARACTERISTICS:
Groups:
- HB-adMSCs: HB-adMSCs (allogeneic)
- Total: Total of all reporting groups
Arm/Group | HB-adMSCs | Placebo | Total
Number analyzed (Participants) | 39 | 40 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 40 | 79
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (10.90) | 42.4 (10.79) | 41.5 (10.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 15 | 36
  Male | 18 | 25 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 18
  Not Hispanic or Latino | 30 | 31 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 38 | 37 | 75
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39 | 40 | 79
Height [Mean (Standard Deviation); unit: centimeter] | 170.76 (7.917) | 174.62 (9,992) | 172.71 (9.177)
Weight [Mean (Standard Deviation); unit: kilograms] | 79.35 (19.229) | 79.28 (15.197) | 79.32 (17.193)

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline in Visual Analog Scale of Neurological Symptoms. - Extreme Fatigue (ANCOVA Model)
Description: Clinically significant changes in Visual Analog Scale - Extreme fatigue. A VAS is a straight line with two end points that represent the extremes of a range. This VAS used to measure extreme fatigue has one end labeled "no fatigue" and the other end labeled "worst fatigue". The patient then marks a point on the line to indicate their current level of fatigue. The minimum score is a 0 and the maximum score is a 10. A higher score indicates a worse outcome (fatigue).
Time Frame: Baseline to Weeks 26
Measure: Mean (Standard Error); unit: score on a scale (10 points total)
Groups:
- HB-adMSCs: HB-adMSCs (allogeneic): HB-adMSCs allogeneic
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
score on a scale (10 points total) | -2.376 (0.496) | -2.430 (0.529)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; The null hypothesis is that the difference in change from baseline to Weeks 26 in Visual Analog Scale of Neurological Symptoms - Extreme fatigue scale score between treatment groups (HB-adMSCs - Placebo) is equal to zero; Test type: Superiority; p = 0.9416, ANCOVA; LS Means = 0.054, 95% CI 2-sided [-1.42 to 1.53], Standard Error of Mean 0.738 — The value described represents the difference value of the mean change from baseline between HB-adMSC and Placebo groups

2. Primary Outcome: Changes From Baseline in Visual Analog Scale of Neurological Symptoms.. - Brain Fog (ANCOVA Model)
Description: Clinically significant changes in Visual Analog Scale - Brain fog. A VAS is a straight line with two end points that represent the extremes of a range. This VAS used to measure brain fog has one end labeled "no brain fog" and the other end labeled "worst brain fog". The patient then marks a point on the line to indicate their current level of brain fog. The minimum score is a 0 and the maximum score is a 10. A higher score indicates a worse outcome (brain fog).
Time Frame: Baseline to Weeks 26
Measure: Mean (Standard Error); unit: score on a scale (10 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
score on a scale (10 points total) | -1.908 (0.462) | -1.736 (0.493)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; The null hypothesis is that the difference in change from baseline to Weeks 26 in Visual Analog Scale of Neurological Symptoms - Brain fog scale score between treatment groups (HB-adMSCs - Placebo) is equal to zero; Test type: Superiority; p = 0.8021, ANCOVA; LS Means = -0.172, 95% CI 2-sided [-1.54 to 1.20], Standard Error of Mean 0.685 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Changes From Baseline in Visual Analog Scale of Neurological Symptoms. - Headache (ANCOVA Model)
Description: Clinically significant changes in Visual Analog Scale - Headache. A VAS is a straight line with two end points that represent the extremes of a range. This VAS used to measure Headache has one end labeled "no headache" and the other end labeled "worst headache". The patient then marks a point on the line to indicate their current level of Headache. The minimum score is a 0 and the maximum score is a 10. A higher score indicates a worse outcome (headache).
Time Frame: Baseline to Weeks 26
Measure: Mean (Standard Error); unit: score on a scale (10 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
score on a scale (10 points total) | -0.755 (0.348) | -1.154 (0.371)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; The null hypothesis is that the difference in change from baseline to Weeks 26 in Visual Analog Scale of Neurological Symptoms. - Headache scale score between treatment groups (HB-adMSCs - Placebo) is equal to zero; Test type: Superiority; p = 0.4417, ANCOVA; LS Means = 0.399, 95% CI 2-sided [-0.63 to 1.43], Standard Error of Mean 0.515 — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Changes From Baseline in Visual Analog Scale of Neurological Symptoms. - Sleep Disturbances (ANCOVA Model)
Description: Clinically significant changes in Visual Analog Scale - Sleep disturbances. A VAS is a straight line with two end points that represent the extremes of a range. This VAS used to measure sleep disturbance has one end labeled "no sleep disturbance" and the other end labeled "worst sleep disturbance". The patient then marks a point on the line to indicate their current level of sleep disturbance. The minimum score is a 0 and the maximum score is a 10. A higher score indicates a worse outcome (sleep disturbance).
Time Frame: Baseline to Weeks 26
Measure: Mean (Standard Error); unit: score on a scale (10 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
score on a scale (10 points total) | -2.005 (0.486) | -2.547 (0.518)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; The null hypothesis is that the difference in change from baseline to Weeks 26 in Visual Analog Scale of Neurological Symptoms - Sleep disturbances scale score between treatment groups (HB-adMSCs - Placebo) is equal to zero; Test type: Superiority; p = 0.4550, ANCOVA; Slope = 0.542, 95% CI 2-sided [-0.90 to 1.98], Standard Error of Mean 0.721

5. Primary Outcome: Changes From Baseline in Visual Analog Scale of Neurological Symptoms. - Loss of Taste (ANCOVA Model)
Description: Clinically significant changes in Visual Analog Scale - Loss of taste. A VAS is a straight line with two end points that represent the extremes of a range. This VAS used to measure loss of taste has one end labeled "no loss of taste" and the other end labeled "worst loss of taste". The patient then marks a point on the line to indicate their current level of loss of taste. The minimum score is a 0 and the maximum score is a 10. A higher score indicates a worse outcome (loss of taste).
Time Frame: Baseline to Weeks 26
Measure: Mean (Standard Error); unit: score on a scale (10 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
score on a scale (10 points total) | -0.509 (0.314) | -0.462 (0.335)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; The null hypothesis is that the difference in change from baseline to Weeks 26 in Visual Analog Scale of Neurological Symptoms - Loss of taste scale score between treatment groups (HB-adMSCs - Placebo) is equal to zero; Test type: Superiority; p = 0.9200, ANCOVA; LS Means = -0.047, 95% CI 2-sided [-0.98 to 0.89], Standard Error of Mean 0.466 — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: Changes From Baseline in Visual Analog Scale of Neurological Symptoms. - Loss of Smell (ANCOVA Model)
Description: Clinically significant changes in Visual Analog Scale - Loss of smell. A VAS is a straight line with two end points that represent the extremes of a range. This VAS used to measure loss of smell has one end labeled "no loss of smell" and the other end labeled "worst loss of smell". The patient then marks a point on the line to indicate their current level of loss of smell. The minimum score is a 0 and the maximum score is a 10. A higher score indicates a worse outcome (loss of smell).
Time Frame: Baseline to Weeks 26
Measure: Mean (Standard Error); unit: score on a scale (10 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
score on a scale (10 points total) | -0.623 (0.241) | -0.463 (0.258)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; The null hypothesis is that the difference in change from baseline to Weeks 26 in PHQ-9 scale score between treatment groups (HB-adMSCs - Placebo) is equal to zero; Test type: Superiority; p = 0.6589, ANCOVA; LS Means = -0.160, 95% CI 2-sided [-0.88 to 0.56], Standard Error of Mean 0.360 — [estimate comment as in outcome 1, analysis 1]

7. Primary Outcome: Changes From Baseline in Visual Analog Scale of Neurological Symptoms - Extreme Fatigue (RMA Model)
Description: Clinically significant changes in Visual Analog Scale. A VAS is a straight line with two end points that represent the extremes of a range. This VAS used to measure extreme fatigue has one end labeled "no fatigue" and the other end labeled "worst fatigue". The patient then marks a point on the line to indicate their current level of fatigue. The minimum score is a 0 and the maximum score is a 10. A higher score indicates a worse outcome (fatigue).
Time Frame: Baseline to Week 26
Measure: Mean (Standard Error); unit: score on a scale (10 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
score on a scale (10 points total)
  Infusion 2 (Week 2) | -1.010 (0.406) | -0.772 (0.428)
  Infusion 3 (Week 6) | -1.214 (0.438) | -1.439 (0.468)
  Infusion 4 (Week 10) | -2.010 (0.463) | -2.018 (0.494)
  EOS (Week 26) | -2.330 (0.490) | -2.492 (0.522)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; The null hypothesis is that the difference in change from baseline to Weeks 26 in Visual Analog Scale of Neurological Symptoms Extreme Fatigue scale score between treatment groups (HB-adMSCs - Placebo) is equal to zero; Test type: Superiority; p = 0.8240, RMA; LS Means = 0.162, 95% CI 2-sided [-1.29 to 1.61], Standard Error of Mean 0.725 — [estimate comment as in outcome 1, analysis 1]

8. Primary Outcome: Changes From Baseline in Visual Analog Scale of Neurological Symptoms.. - Brain Fog (RMA Model)
Description: as for outcome 2
Time Frame: Baseline to Week 26
Measure: Mean (Standard Error); unit: score on a scale (10 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
score on a scale (10 points total)
  Infusion 2 (Week 2) | -1.134 (0.352) | -0.944 (0.371)
  Infusion 3 (Week 6) | -1.425 (0.377) | -0.837 (0.402)
  Infusion 4 (Week 10) | -2.281 (0.419) | -1.532 (0.446)
  End of Study (Week 26) | -1.827 (0.467) | -1.818 (0.497)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.9892, RMA; LS Means = -0.009, 95% CI 2-sided [-1.38 to 1.36], Standard Error of Mean 0.686 — [estimate comment as in outcome 1, analysis 1]

9. Primary Outcome: Changes From Baseline in Visual Analog Scale of Neurological Symptoms. - Headache (RMA Model)
Description: as for outcome 3
Time Frame: Baseline to Week 26
Measure: Mean (Standard Error); unit: score on a scale (10 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
score on a scale (10 points total)
  Infusion 2 (Week 2) | -0.362 (0.400) | -0.548 (0.422)
  Infusion 3 (Week 6) | -0.504 (0.388) | -0.648 (0.414)
  Infusion 4 (Week 10) | -0.696 (0.385) | -0.870 (0.411)
  End Of Study (Week 26) | -0.741 (0.346) | -1.181 (0.369)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; The null hypothesis is that the difference in change from baseline to Weeks 26 in Visual Analog Scale of Neurological Symptoms - Headache scale score between treatment groups (HB-adMSCs - Placebo) is equal to zero; Test type: Superiority; p = 0.3952, RMA; LS Means = 0.439, 95% CI 2-sided [-0.59 to 1.47], Standard Error of Mean 0.513 — [estimate comment as in outcome 1, analysis 1]

10. Primary Outcome: Changes From Baseline in Visual Analog Scale of Neurological Symptoms. - Sleep Disturbances (RMA Model)
Description: as for outcome 4
Time Frame: Baseline to Weeks 26
Measure: Mean (Standard Error); unit: score on a scale (10 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
score on a scale (10 points total)
  Infusion 2 (Week 2) | -1.331 (0.340) | -0.730 (0.357)
  Infusion 3 (Week 6) | -1.845 (0.462) | -1.813 (0.492)
  Infusion 4 (Week 10) | -2.028 (0.466) | -2.095 (0.497)
  End of Study (Week 26) | -2.016 (0.479) | -2.551 (0.510)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.4504, RMA; LS Means = 0.535, 95% CI 2-sided [-0.87 to 1.94], Standard Error of Mean 0.704 — [estimate comment as in outcome 1, analysis 1]

11. Primary Outcome: Changes From Baseline in Visual Analog Scale of Neurological Symptoms. - Loss of Taste (RMA Model)
Description: as for outcome 5
Time Frame: Baseline to Weeks 26
Measure: Mean (Standard Error); unit: score on a scale (10 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
score on a scale (10 points total)
  Infusion 2 (Week 2) | -0.450 (0.234) | 0.235 (0.247)
  Infusion 3 (Week 6) | -0.372 (0.325) | 0.523 (0.346)
  Infusion 4 (Week 10) | -0.654 (0.339) | -0.365 (0.362)
  End of Study (Week 26) | -0.569 (0.318) | -0.408 (0.339)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.7318, RMA; LS Means = -0.161, 95% CI 2-sided [-1.10 to 0.78], Standard Error of Mean 0.469 — [estimate comment as in outcome 1, analysis 1]

12. Primary Outcome: Changes From Baseline in Visual Analog Scale of Neurological Symptoms. - Loss of Smell (RMA Model)
Description: as for outcome 6
Time Frame: Baseline to Weeks 26
Measure: Mean (Standard Error); unit: score on a scale (10 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
score on a scale (10 points total)
  Infusion 2 (Week 2) | -0.336 (0.273) | 0.617 (0.288)
  Infusion 3 (Week 6) | -0.112 (0.264) | -0.013 (0.281)
  Infusion 4 (Week 10) | -0.678 (0.242) | -0.196 (0.258)
  End Of Study (Week 26) | -0.653 (0.241) | -0.438 (0.256)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; The null hypothesis is that the difference in change from baseline to Weeks 26 in Visual Analog Scale of Neurological Symptoms - Loss of Smell scale score between treatment groups (HB-adMSCs - Placebo) is equal to zero; Test type: Superiority; p = 0.5485, RMA; LS Means = -0.215, 95% CI 2-sided [-0.93 to 0.50], Standard Error of Mean 0.357 — [estimate comment as in outcome 1, analysis 1]

13. Primary Outcome: Changes in Laboratory Values. - CBC. (x10^3 Cells/uL)
Description: Clinically significant changes in CBC values.
Time Frame: Baseline to Weeks 26
Measure: Mean (Standard Error); unit: x10^3 cells/uL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
x10^3 cells/uL
  Absolute Basophils Baseline/Infusion 1 (Week 0) | 0.0454 (0.00531) | 0.0415 (0.00315)
  Absolute Basophils Infusion 4 (Week 10) | 0.0017 (0.00344) | 0.0047 (0.00327)
  Absolute Basophils End of Study (Week 26) | -0.0019 (0.00407) | 0.0037 (0.00344)
  Absolute Eosinophils Baseline/Infusion 1 (Week 0) | 0.1177 (0.01258) | 0.1965 (0.03371)
  Absolute Eosinophils Infusion 4 (Week 10) | 0.0006 (0.00903) | -0.0356 (0.02410)
  Absolute Eosinophils End of Study (Week 26) | 0.0105 (0.01051) | -0.0373 (0.03355)
  Absolute Lymphocytes Baseline/Infusion 1 (Week 0) | 1.9733 (0.10847) | 1.8820 (0.09517)
  Absolute Lymphocytes Infusion 4 (Week 10) | -0.0623 (0.07443) | -0.0203 (0.06454)
  Absolute Lymphocytes End of Study (Week 26) | 0.0851 (0.09160) | -0.0777 (0.07055)
  Absolute Monocytes Baseline/Infusion 1 (Week 0) | 0.4877 (0.02321) | 0.4663 (0.01919)
  Absolute Monocytes Infusion 4 (Week 10) | -0.0269 (0.02181) | 0.0084 (0.01992)
  Absolute Monocytes End of Study (Week 26) | 0.0324 (0.02022) | -0.0040 (0.01791)
  Absolute Neutrophils Baseline/Infusion 1 (Week 0) | 3.4426 (0.18489) | 3.2103 (0.16672)
  Absolute Neutrophils Infusion 4 (Week 10) | 0.0900 (0.29868) | 0.0591 (0.15940)
  Absolute Neutrophils End of Study (Week 26) | 0.1785 (0.19430) | 0.0883 (0.15998)
  Platelet Baseline/Infusion 1 (Week 0) | 269.1 (8.73) | 249.4 (8.25)
  Platelet Infusion 4 (Week 10) | -11.9 (5.77) | 2.3 (6.18)
  Platelet End of Study (Week 26) | -2.1 (5.37) | 2.1 (5.94)
  WBC Baseline/Infusion 1 (Week 0) | 6.08 (0.279) | 5.82 (0.255)
  WBC Infusion 4 (Week 10) | 0.01 (0.311) | 0.02 (0.188)
  WBC End of Study (Week 26) | 0.30 (0.261) | -0.04 (0.183)

14. Primary Outcome: Changes in Laboratory Values. - CBC. (% of WBC)
Description: Clinically significant changes in CBC values.
Time Frame: Baseline to Weeks 26
Measure: Mean (Standard Error); unit: % of WBC
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
% of WBC
  Basophils Baseline/Infusion 1 (Week 0) | 0.91 (0.135) | 1.07 (0.168)
  Basophils Infusion 4 (Week 10) | -0.21 (0.144) | -0.08 (0.188)
  Basophils End of Study (Week 26) | -0.08 (0.197) | 0.02 (0.136)
  Eosinophils Baseline/Infusion 1 (Week 0) | 1.99 (0.252) | 3.00 (0.468)
  Eosinophils Infusion 4 (Week 10) | -0.11 (0.243) | -0.52 (0.461)
  Eosinophils End of Study (Week 26) | 0.26 (0.326) | -0.41 (0.421)
  Lymphocytes Baseline/Infusion 1 (Week 0) | 34.29 (1.213) | 36.20 (1.239)
  Lymphocytes Infusion 4 (Week 10) | -0.49 (1.662) | -1.46 (1.548)
  Lymphocytes End of Study (Week 26) | -0.56 (1.379) | -3.25 (1.444)
  Monocytes Baseline/Infusion 1 (Week 0) | 7.79 (0.545) | 7.27 (0.382)
  Monocytes Infusion 4 (Week 10) | -0.29 (0.426) | 0.61 (0.583)
  Monocytes End of Study (Week 26) | 0.24 (0.642) | 0.54 (0.472)
  Neutrophils Baseline/Infusion 1 (Week 0) | 54.95 (1.162) | 52.37 (1.508)
  Neutrophils Infusion 4 (Week 10) | 1.05 (1.850) | 1.44 (2.131)
  Neutrophils End of Study (Week 26) | 0.06 (1.681) | 3.03 (1.675)

15. Primary Outcome: Changes in Laboratory Values. - CBC (pg)
Description: Changes from baseline in CBC laboratory values with unit of pg.
Time Frame: Baseline (Week 0), Week 10, and End of Study (Week 26)
Measure: Mean (Standard Error); unit: pg
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
pg
  MCH Baseline/Infusion 1 (Week 0) | 30.40 (0.242) | 30.64 (0.226)
  MCH Infusion 4 (Week 10) | -0.00 (0.134) | -0.06 (0.133)
  MCH End of Study (Week 26) | -0.06 (0.169) | -0.14 (0.201)

16. Primary Outcome: Changes in Laboratory Values. - CBC (g/dL)
Description: Changes from baseline in CBC laboratory values with unit of g/dL.
Time Frame: Baseline (Week 0), Week 10, and End of Study (Week 26)
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
g/dL
  MCHC Baseline/Infusion 1 (Week 0) | 33.90 (0.155) | 34.05 (0.138)
  MCHC Infusion 4 (Week 10) | -0.05 (0.143) | 0.04 (0.185)
  MCHC End of Study (Week 26) | -0.24 (0.160) | -0.23 (0.245)
  Hemoglobin Baseline/Infusion 1 (Week 0) | 14.35 (0.235) | 14.34 (0.211)
  Hemoglobin Infusion 4 (Week 10) | -0.11 (0.133) | 0.13 (0.102)
  Hemoglobin End of Study (Week 26) | -0.13 (0.131) | 0.13 (0.158)

17. Primary Outcome: Changes in Laboratory Values. - CBC (fL)
Description: Changes from baseline in CBC laboratory values with unit of fL.
Time Frame: Baseline (Week 0), Week 10, and End of Study (Week 26)
Measure: Mean (Standard Error); unit: fL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
fL
  MCV Baseline/Infusion 1 (Week 0) | 89.68 (0.575) | 90.00 (0.485)
  MCV Infusion 4 (Week 10) | 0.14 (0.204) | -0.29 (0.327)
  MCV End of Study (Week 26) | 0.42 (0.350) | 0.21 (0.318)

18. Primary Outcome: Changes in Laboratory Values. - CBC (x10^6 Cells/uL)
Description: Changes from baseline in CBC laboratory values with unit of 10^6 cells/uL.
Time Frame: Baseline (Week 0), Week 10, and End of Study (Week 26)
Measure: Mean (Standard Error); unit: 10^6 cells/uL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
10^6 cells/uL
  RBC Baseline/Infusion 1 (Week 0) | 4.729 (0.0822) | 4.690 (0.0804)
  RBC Infusion 4 (Week 10) | -0.039 (0.0460) | 0.052 (0.0384)
  RBC End of Study (Week 26) | -0.033 (0.0507) | 0.062 (0.0547)

19. Primary Outcome: Changes in Laboratory Values. - CBC (% Difference in Volume and Size of RBC)
Description: Changes from baseline in CBC laboratory values with unit % Difference in Volume and Size of RBC
Time Frame: Baseline (Week 0), Week 10, and End of Study (Week 26)
Measure: Mean (Standard Error); unit: % difference in volume and size of RBC
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
% difference in volume and size of RBC
  RDW Baseline/Infusion 1 (Week 0) | 12.58 (0.107) | 12.58 (0.104)
  RDW Infusion 4 (Week 10) | -0.03 (0.071) | -0.08 (0.100)
  RDW End of Study (Week 26) | 0.01 (0.096) | 0.01 (0.060)

20. Primary Outcome: Changes in Laboratory Values. - CBC (% of Total Blood Cell Count)
Description: Changes from baseline in CBC laboratory values with unit of % of Total Blood Cell Count.
Time Frame: Baseline (Week 0), Week 10, and End of Study (Week 26)
Measure: Mean (Standard Error); unit: % of Total Blood Cell Count
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
% of Total Blood Cell Count
  Hematocrit Baseline/Infusion 1 (Week 0) | 42.33 (0.652) | 42.11 (0.600)
  Hematocrit Infusion 4 (Week 10) | -0.27 (0.405) | 0.32 (0.336)
  Hematocrit End of Study (Week 26) | -0.11 (0.444) | 0.64 (0.443)

21. Primary Outcome: Changes in Laboratory Values. - CMP (g/dL)
Description: Clinically significant changes in CMP values.
Time Frame: Baseline (Week 0), Week 10, and End of Study (Week 26)
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
g/dL
  Albumin Baseline/Infusion 1 (Week 0) | 4.65 (0.052) | 4.63 (0.045)
  Albumin Infusion 4 (Week 10) | -0.11 (0.039) | -0.02 (0.044)
  Albumin End of Study (Week 26) | -0.13 (0.039) | -0.02 (0.052)
  Calc Globulin Baseline/Infusion 1 (Week 0) | 2.63 (0.125) | 2.46 (0.063)
  Calc Globulin Infusion 4 (Week 10) | -0.08 (0.045) | 0.03 (0.043)
  Calc Globulin End of Study (Week 26) | -0.07 (0.061) | -0.05 (0.047)
  Protein Baseline/Infusion 1 (Week 0) | 7.28 (0.113) | 7.09 (0.068)
  Protein Infusion 4 (Week 10) | -0.19 (0.068) | 0.02 (0.057)
  Protein End of Study (Week 26) | -0.20 (0.072) | -0.07 (0.075)

22. Primary Outcome: Changes in Laboratory Values. - Coagulation Panel. Ratio: Prothrombin Time (Seconds) / Mean Normal Prothrombin Time (Seconds
Description: Clinically significant changes in Coagulation Panel values with units of Ratio: Prothrombin time (seconds) / Mean normal prothrombin time (seconds).
Time Frame: Baseline (Week 0), Week 10, and End of Study (Week 26)
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
Ratio
  INR Baseline/Infusion 1 (Week 0) | 0.99 (0.010) | 0.97 (0.011)
  INR Infusion 4 (Week 10) | -0.01 (0.008) | 0.01 (0.010)
  INR End of Study (Week 26) | 0.00 (0.011) | -0.01 (0.013)

23. Primary Outcome: Changes From Baseline in Vital Signs. - Respiratory Rate (Breaths Per Minute)
Description: Clinically significant changes in Respiratory Rate (breaths per minute)
Time Frame: Baseline to Weeks 26
Measure: Mean (Standard Error); unit: breaths/min
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
breaths/min
  Baseline | 17.0 (0.16) | 16.8 (0.16)
  Infusion 2 (Week 2) | 0.1 (0.19) | 0.2 (0.22)
  Infusion 3 (Week 6) | -0.1 (0.21) | 0.2 (0.19)
  Infusion 4 (Week 10) | -0.3 (0.15) | -0.1 (0.22)
  End of Study (Week 26) | 0.1 (0.20) | 0.3 (0.24)

24. Primary Outcome: Changes From Baseline in Vital Signs. - Heart Rate (Beats Per Minute)
Description: Clinically significant changes in Heart Rate (beats per minute)
Time Frame: Baseline to Weeks 26
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
beats per minute
  Baseline | 73.9 (1.88) | 70.0 (1.76)
  Infusion 2 (Week 2) | -0.6 (1.67) | 3.6 (1.65)
  Infusion 3 (Week 6) | 0.5 (2.07) | 6.1 (2.14)
  Infusion 4 (Week 10) | -3.5 (1.91) | 3.2 (1.65)
  End of Study (Week 26) | -4.2 (2.09) | 2.4 (1.54)

25. Primary Outcome: Changes From Baseline in Vital Signs. - Body Temperature (Celsius)
Description: Clinically significant changes in Body Temperature (Celsius)
Time Frame: Baseline to Week 10, End of Study at Weeks 26
Measure: Mean (Standard Error); unit: degrees Celsius
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
degrees Celsius
  Baseline | 36.63 (0.043) | 36.70 (0.039)
  Infusion 2 (Week 2) | 0.01 (0.047) | -0.04 (0.040)
  Infusion 3 (Week 6) | 0.05 (0.050) | -0.03 (0.050)
  Infusion 4 (Week 10) | 0.01 (0.051) | -0.05 (0.038)
  End of Study (Week 26) | -0.08 (0.052) | -0.05 (0.053)

26. Primary Outcome: Changes in Vital Signs. - Blood Pressure (mmHg)
Description: Clinically significant changes in Blood Pressure.
Time Frame: Baseline to Weeks 10, End of Study at Week 26
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
mmHg
  Systolic Basline/Infusion 1 (Week 0) | 122.2 (1.91) | 125.2 (1.78)
  Systolic Infusion 2 (Week 2) | -0.7 (1.82) | -1.8 (1.51)
  Systolic Infusion 3 (Week 6) | -0.6 (1.85) | 1.1 (1.57)
  Systolic Infusion 4 (Week 10) | -3.1 (2.10) | -3.1 (1.52)
  Systolic End of Study (Week 26) | -0.2 (1.74) | 0.3 (1.78)
  Diastolic Baseline/Infusion 1 (Week 0) | 79.4 (1.32) | 80.1 (1.06)
  Diastolic Infusion 2 (Week 2) | -0.9 (0.98) | -0.7 (0.92)
  Diastolic Infusion 3 (Week 6) | -2.2 (1.48) | 0.1 (1.31)
  Diastolic Infusion 4 (Week 10) | -0.8 (1.50) | -0.6 (1.46)
  Diastolic End of Study (Week 26) | 0.0 (1.32) | 1.1 (1.39)

27. Primary Outcome: Changes in Weight in kg.
Description: Change from baseline in Weight in kg.
Time Frame: Baseline to Weeks 10, End of Study at Week 26
Measure: Mean (Standard Error); unit: kg
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
kg
  Baseline/ Infusion 1 (Week 0) | 79.35 (3.079) | 79.28 (2.403)
  Infusion 2 (Week 2) | -0.06 (0.342) | 0.80 (0.551)
  Infusion 3 (Week 6) | 0.26 (0.476) | 1.15 (0.602)
  Infusion 4 (Week 10) | 0.49 (0.645) | 0.56 (0.627)
  End of Study (Week 26) | -0.30 (0.751) | 1.14 (0.925)

28. Primary Outcome: Changes in Physical Examination Results. - Abdomen
Description: Clinically significant changes in physical examination results - Abdomen body system
Time Frame: Baseline to Week 10, Follow-up at Week 14, End of Study at Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
Participants
  Baseline/Infusion 1 (Week 0): Normal | 38 | 38
  Baseline/Infusion 1 (Week 0): Abnormal | 1 | 2
  Baseline/Infusion 1 (Week 0): Not Examined (No Longer In Study) | 0 | 0
  Infusion 2 (Week 2): Normal | 37 | 36
  Infusion 2 (Week 2): Abnormal | 0 | 0
  Infusion 2 (Week 2): Not Examined (No Longer In Study) | 2 | 4
  Infusion 3 (Week 6): Normal | 36 | 34
  Infusion 3 (Week 6): Abnormal | 1 | 1
  Infusion 3 (Week 6): Not Examined (No Longer In Study) | 2 | 5
  Infusion 4 (Week 10): Normal | 35 | 32
  Infusion 4 (Week 10): Abnormal | 0 | 0
  Infusion 4 (Week 10): Not Examined (No Longer In Study) | 4 | 8
  End of Study (Week 26): Normal | 34 | 30
  End of Study (Week 26): Abnormal | 0 | 0
  End of Study (Week 26): Not Examined (No Longer In Study) | 5 | 10

29. Primary Outcome: Changes in Laboratory Values. - CMP (Ratio: Albumin (g/dL) to Calc. Globulin (g/dL)
Description: Changes from baseline in CMP laboratory values with units of Ratio: Albumin(g/dL) to Calc. Globulin(g/dL)
Time Frame: Baseline (Week 0), Week 10, and End of Study (Week 26)
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
Ratio
  Calc A/G Ratio Baseline/Infusion 1 (Week 0) | 1.86 (0.057) | 1.94 (0.060)
  Calc A/G Ratio Infusion 4 (Week 10) | 0.02 (0.044) | -0.03 (0.046)
  Calc A/G Ratio End of Study (Week 26) | 0.04 (0.053) | 0.03 (0.043)

30. Primary Outcome: Changes in Laboratory Values. - CMP (U/L)
Description: Clinically significant changes in CMP values with units of U/L.
Time Frame: Baseline (Week 0), Week 10, and End of Study (Week 26)
Measure: Mean (Standard Error); unit: U/L
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
U/L
  Alkaline Phosphatase Baseline/Infusion 1 (Week 0) | 66.9 (2.31) | 74.5 (3.42)
  Alkaline Phosphatase Infusion 4 (Week 10) | -3.2 (1.51) | 0.1 (1.29)
  Alkaline Phosphatase End of Study (Week 26) | -4.1 (1.56) | -0.5 (1.87)
  Alanine aminotransferase Baseline/Infusion 1 (Week 0) | 25.15 (1.836) | 21.28 (1.718)
  Alanine aminotransferase Infusion 4 (Week 10) | -5.14 (1.272) | 2.81 (1.353)
  Alanine aminotransferase End of Study (Week 26) | 0.26 (3.321) | 2.00 (1.211)
  Aspartate Aminotransferase Baseline/Infusion 1 (Week 0) | 23.8 (1.63) | 20.7 (0.96)
  Aspartate Aminotransferase Infusion 4 (Week 10) | -2.9 (1.56) | 1.5 (1.17)
  Aspartate Aminotransferase End of Study (Week 26) | -0.7 (2.25) | 0.6 (1.09)

31. Primary Outcome: Changes in Laboratory Values. - CMP (mg/dL)
Description: Clinically significant changes in CMP values with units of mg/dL.
Time Frame: Baseline (Week 0), Week 10, and End of Study (Week 26)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
mg/dL
  Bilirubin Baseline/Infusion 1 (Week 0) | 0.52 (0.029) | 0.50 (0.043)
  Bilirubin Infusion 4 (Week 10) | -0.05 (0.035) | 0.03 (0.034)
  Bilirubin End of Study (Week 26) | -0.12 (0.032) | -0.01 (0.047)
  Calcium Baseline/Infusion 1 (Week 0) | 9.56 (0.085) | 9.54 (0.055)
  Calcium Infusion 4 (Week 10) | -0.04 (0.099) | -0.01 (0.058)
  Calcium End of Study (Week 26) | -0.06 (0.098) | -0.03 (0.065)
  Creatinine Baseline/Infusion 1 (Week 0) | 0.885 (0.0337) | 0.872 (0.0290)
  Creatinine Infusion 4 (Week 10) | -0.022 (0.0146) | -0.010 (0.0103)
  Creatinine End of Study (Week 26) | -0.012 (0.0190) | 0.014 (0.0106)
  Glucose Baseline/Infusion 1 (Week 0) | 98.5 (6.43) | 94.2 (1.93)
  Glucose Infusion 4 (Week 10) | -5.0 (6.40) | 0.7 (2.35)
  Glucose End of Study (Week 26) | -2.9 (4.92) | 2.0 (1.41)
  Blood Urea Nitrogen Baseline/Infusion 1 (Week 0) | 13.9 (0.61) | 13.8 (0.51)
  Blood Urea Nitrogen Infusion 4 (Week 10) | -0.3 (0.54) | -0.1 (0.64)
  Blood Urea Nitrogen End of Study (Week 26) | 0.4 (0.67) | -0.2 (0.62)

32. Primary Outcome: Changes in Laboratory Values. - CMP (mEq/L)
Description: Clinically significant changes in CMP values with units of mEq/L.
Time Frame: Baseline (Week 0), Week 10, and End of Study (Week 26)
Measure: Mean (Standard Error); unit: mEq/L
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
mEq/L
  Chloride Baseline/Infusion 1 (Week 0) | 103.3 (0.45) | 104.1 (0.35)
  Chloride Infusion 4 (Week 10) | 0.2 (0.45) | -0.3 (0.37)
  Chloride End of Study (Week 26) | 0.6 (0.42) | -0.3 (0.40)
  Carbon Dioxide Baseline/Infusion 1 (Week 0) | 24.7 (0.33) | 25.2 (0.35)
  Carbon Dioxide Infusion 4 (Week 10) | -0.2 (0.39) | -0.3 (0.43)
  Carbon Dioxide End of Study (Week 26) | 0.0 (0.47) | -0.4 (0.45)
  Potassium Baseline/Infusion 1 (Week 0) | 4.40 (0.059) | 4.44 (0.086)
  Potassium Infusion 4 (Week 10) | -0.08 (0.067) | -0.08 (0.128)
  Potassium End of Study (Week 26) | -0.14 (0.080) | -0.11 (0.118)
  Sodium Baseline/Infusion 1 (Week 0) | 140.2 (0.38) | 141.1 (0.31)
  Sodium Infusion 4 (Week 10) | -0.1 (0.45) | 0.2 (0.50)
  Sodium End of Study (Week 26) | 0.2 (0.51) | -0.5 (0.49)

33. Primary Outcome: Changes in Laboratory Values. - CMP (mL/Min/1.73m^2)
Description: Clinically significant changes in CMP values with units of mL/min/1.73m^2.
Time Frame: Baseline (Week 0), Week 10, and End of Study (Week 26)
Measure: Mean (Standard Error); unit: mL/min/1.73m^2
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
mL/min/1.73m^2
  Estimated Glomerular Filtration Rate Baseline/Infusion 1 (Week 0) | 97.6 (2.45) | 101.1 (2.06)
  Estimated Glomerular Filtration Rate Infusion 4 (Week 10) | 1.8 (1.54) | 0.9 (1.10)
  Estimated Glomerular Filtration Rate End of Study (Week 26) | 0.7 (1.88) | -1.2 (1.27)

34. Primary Outcome: Changes in Laboratory Values. - CMP (Calc BUN mg/dL /Creat mg/dL Ratio)
Description: Clinically significant changes in CMP values with units of Calc BUN mg/dL /Creat mg/dL Ratio
Time Frame: Baseline (Week 0), Week 10, and End of Study (Week 26)
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
Ratio
  Calc BUN/Creat Baseline/Infusion 1 (Week 0) | 16.5 (0.97) | 16.4 (0.68)
  Calc BUN/Creat Infusion 4 (Week 10) | -0.0 (0.64) | -0.1 (0.68)
  Calc BUN/Creat End of Study (Week 26) | 0.7 (0.82) | -0.4 (0.75)

35. Primary Outcome: Changes in Laboratory Values. - Coagulation Panel. (Seconds)
Description: Clinically significant changes in Coagulation Panel values with units of seconds.
Time Frame: Baseline (Week 0), Week 10, and End of Study (Week 26)
Measure: Mean (Standard Error); unit: seconds
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
seconds
  Prothrombin Time Baseline/Infusion 1 (Week 0) | 13.42 (0.092) | 13.27 (0.097)
  Prothrombin Time Infusion 4 (Week 10) | -0.11 (0.057) | 0.05 (0.081)
  Prothrombin Time End of Study (Week 26) | -0.12 (0.115) | -0.05 (0.085)
  PTT Baseline/Infusion 1 (Week 0) | 29.36 (0.486) | 29.93 (0.416)
  PTT Infusion 4 (Week 10) | -0.54 (0.302) | -0.51 (0.198)
  PTT End of Study (Week 26) | -0.48 (0.261) | -0.73 (0.238)

36. Primary Outcome: Changes in Physical Examination Results. - Cardiovascular
Description: Clinically significant changes in physical examination results - Cardiovascular body system
Time Frame: Baseline to Week 10, Follow-up at Week 14, End of Study at Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
Participants
  Baseline/Infusion 1 (Week 0): Normal | 38 | 39
  Baseline/Infusion 1 (Week 0): Abnormal | 1 | 1
  Baseline/Infusion 1 (Week 0): Not Examined (No Longer In Study) | 0 | 0
  Infusion 2 (Week 2): Normal | 37 | 36
  Infusion 2 (Week 2): Abnormal | 0 | 0
  Infusion 2 (Week 2): Not Examined (No Longer In Study) | 2 | 4
  Infusion 3 (Week 6): Normal | 37 | 33
  Infusion 3 (Week 6): Abnormal | 0 | 2
  Infusion 3 (Week 6): Not Examined (No Longer In Study) | 2 | 5
  Infusion 4 (Week 10): Normal | 35 | 32
  Infusion 4 (Week 10): Abnormal | 0 | 0
  Infusion 4 (Week 10): Not Examined (No Longer In Study) | 4 | 8
  End of Study (Week 26): Normal | 34 | 30
  End of Study (Week 26): Abnormal | 0 | 0
  End of Study (Week 26): Not Examined (No Longer In Study) | 5 | 10

37. Primary Outcome: Changes in Physical Examination Results. - Head, Eyes, Ears, Nose, and Throat
Description: Clinically significant changes in physical examination results - Head, Eyes, Ears, Nose, and Throat body system
Time Frame: Baseline to Week 10, Follow-up at Week 14, End of Study at Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
Participants
  Baseline/Infusion 1 (Week 0): Normal | 39 | 40
  Baseline/Infusion 1 (Week 0): Abnormal | 0 | 0
  Baseline/Infusion 1 (Week 0): Not Examined (No Longer In Study) | 0 | 0
  Infusion 2 (Week 2): Normal | 37 | 36
  Infusion 2 (Week 2): Abnormal | 0 | 0
  Infusion 2 (Week 2): Not Examined (No Longer In Study) | 2 | 4
  Infusion 3 (Week 6): Normal | 36 | 35
  Infusion 3 (Week 6): Abnormal | 1 | 0
  Infusion 3 (Week 6): Not Examined (No Longer In Study) | 2 | 5
  Infusion 4 (Week 10): Normal | 35 | 32
  Infusion 4 (Week 10): Abnormal | 0 | 0
  Infusion 4 (Week 10): Not Examined (No Longer In Study) | 4 | 8
  End of Study (Week 26): Normal | 34 | 30
  End of Study (Week 26): Abnormal | 0 | 0
  End of Study (Week 26): Not Examined (No Longer In Study) | 5 | 10

38. Primary Outcome: Changes in Physical Examination Results. - Lymph Node
Description: Clinically significant changes in physical examination results - Lymph Node
Time Frame: Baseline to Week 10, Follow-up at Week 14, End of Study at Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
Participants
  Baseline/Infusion 1 (Week 0): Normal | 39 | 40
  Baseline/Infusion 1 (Week 0): Abnormal | 0 | 0
  Baseline/Infusion 1 (Week 0): Not Examined (No Longer In Study) | 0 | 0
  Infusion 2 (Week 2): Normal | 37 | 36
  Infusion 2 (Week 2): Abnormal | 0 | 0
  Infusion 2 (Week 2): Not Examined (No Longer In Study) | 2 | 4
  Infusion 3 (Week 6): Normal | 37 | 35
  Infusion 3 (Week 6): Abnormal | 0 | 0
  Infusion 3 (Week 6): Not Examined (No Longer In Study) | 2 | 5
  Infusion 4 (Week 10): Normal | 35 | 32
  Infusion 4 (Week 10): Abnormal | 0 | 0
  Infusion 4 (Week 10): Not Examined (No Longer In Study) | 4 | 8
  End of Study (Week 26): Normal | 34 | 30
  End of Study (Week 26): Abnormal | 0 | 0
  End of Study (Week 26): Not Examined (No Longer In Study) | 5 | 10

39. Primary Outcome: Changes in Physical Examination Results. - Musculoskeletal
Description: Clinically significant changes in physical examination results - Musculoskeletal
Time Frame: Baseline to Week 10, Follow-up at Week 14, End of Study at Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
Participants
  Baseline/Infusion 1 (Week 0): Normal | 37 | 40
  Baseline/Infusion 1 (Week 0): Abnormal | 2 | 0
  Baseline/Infusion 1 (Week 0): Not Examined (No Longer In Study) | 0 | 0
  Infusion 2 (Week 2): Normal | 35 | 35
  Infusion 2 (Week 2): Abnormal | 2 | 1
  Infusion 2 (Week 2): Not Examined (No Longer In Study) | 2 | 4
  Infusion 3 (Week 6): Normal | 35 | 34
  Infusion 3 (Week 6): Abnormal | 2 | 1
  Infusion 3 (Week 6): Not Examined (No Longer In Study) | 2 | 5
  Infusion 4 (Week 10): Normal | 34 | 32
  Infusion 4 (Week 10): Abnormal | 1 | 0
  Infusion 4 (Week 10): Not Examined (No Longer In Study) | 4 | 8
  End of Study (Week 26): Normal | 33 | 30
  End of Study (Week 26): Abnormal | 1 | 0
  End of Study (Week 26): Not Examined (No Longer In Study) | 5 | 10

40. Primary Outcome: Changes in Physical Examination Results. - Neurological
Description: Clinically significant changes in physical examination results - Neurological
Time Frame: Baseline to Week 10, Follow-up at Week 14, End of Study at Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
Participants
  Baseline/ Infusion 1: Normal | 30 | 39
  Baseline/ Infusion 1: Abnormal | 9 | 1
  Baseline/ Infusion 1: Not Examined (No Longer In Study) | 0 | 0
  Infusion 2 (Week 2): Normal | 35 | 36
  Infusion 2 (Week 2): Abnormal | 2 | 0
  Infusion 2 (Week 2): Not Examined (No Longer In Study) | 2 | 4
  Infusion 3 (Week 6): Normal | 32 | 35
  Infusion 3 (Week 6): Abnormal | 5 | 0
  Infusion 3 (Week 6): Not Examined (No Longer In Study) | 2 | 5
  Infusion 4 (Week 10): Normal | 31 | 31
  Infusion 4 (Week 10): Abnormal | 4 | 1
  Infusion 4 (Week 10): Not Examined (No Longer In Study) | 4 | 8
  End of Study (Week 26): Normal | 31 | 30
  End of Study (Week 26): Abnormal | 3 | 0
  End of Study (Week 26): Not Examined (No Longer In Study) | 5 | 10

41. Primary Outcome: Changes in Physical Examination Results. - Respiratory
Description: Clinically significant changes in physical examination results - Respiratory
Time Frame: Baseline to Week 10, Follow-up at Week 14, End of Study at Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
Participants
  Baseline/Infusion 1 (Week 0): Normal | 38 | 39
  Baseline/Infusion 1 (Week 0): Abnormal | 1 | 1
  Baseline/Infusion 1 (Week 0): Not Examined (No Longer In Study) | 0 | 0
  Infusion 2 (Week 2): Normal | 37 | 36
  Infusion 2 (Week 2): Abnormal | 0 | 0
  Infusion 2 (Week 2): Not Examined (No Longer In Study) | 2 | 4
  Infusion 3 (Week 6): Normal | 37 | 35
  Infusion 3 (Week 6): Abnormal | 0 | 0
  Infusion 3 (Week 6): Not Examined (No Longer In Study) | 2 | 5
  Infusion 4 (Week 10): Normal | 35 | 31
  Infusion 4 (Week 10): Abnormal | 0 | 1
  Infusion 4 (Week 10): Not Examined (No Longer In Study) | 4 | 8
  End of Study (Week 26): Normal | 34 | 29
  End of Study (Week 26): Abnormal | 0 | 1
  End of Study (Week 26): Not Examined (No Longer In Study) | 5 | 10

42. Primary Outcome: Changes in Physical Examination Results. - Skin
Description: Clinically significant changes in physical examination results - Skin. Patients are ranked as normal or abnormal per body system.
Time Frame: Baseline to Week 10, Follow-up at Week 14, End of Study at Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
Participants
  Baseline/Infusion 1 (Week 0): Normal | 39 | 39
  Baseline/Infusion 1 (Week 0): Abnormal | 0 | 1
  Baseline/Infusion 1 (Week 0): Not Examined (No Longer In Study) | 0 | 0
  Infusion 2 (Week 2): Normal | 35 | 34
  Infusion 2 (Week 2): Abnormal | 2 | 2
  Infusion 2 (Week 2): Not Examined (No Longer In Study) | 2 | 4
  Infusion 3 (Week 6): Normal | 37 | 34
  Infusion 3 (Week 6): Abnormal | 0 | 1
  Infusion 3 (Week 6): Not Examined (No Longer In Study) | 2 | 5
  Infusion 4 (Week 10): Normal | 34 | 31
  Infusion 4 (Week 10): Abnormal | 1 | 1
  Infusion 4 (Week 10): Not Examined (No Longer In Study) | 4 | 8
  End of Study (Week 26): Normal | 34 | 30
  End of Study (Week 26): Abnormal | 0 | 0
  End of Study (Week 26): Not Examined (No Longer In Study) | 5 | 10

43. Secondary Outcome: Changes From Baseline in Visual Analog Scale of Non-Neurological Symptoms. - Dyspnea at Rest (ANCOVA Model)
Description: Clinically significant changes in Visual Analog Scale - Dyspnea at rest. Score ranges from 0 points (no dyspnea) to 10 points (maximum amount of dyspnea).
Time Frame: Baseline (Infusion 1) to Weeks 26 (End of Study)
Measure: Mean (Standard Error); unit: score on a scale (10 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
score on a scale (10 points total) | -1.354 (0.275) | -0.976 (0.293)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; The null hypothesis is that the difference in change from baseline to Weeks 26 in Visual Analog Scale of Non-Neurological Symptoms. - Dyspnea at rest scale score between treatment groups (HB-adMSCs - Placebo) is equal to zero; Test type: Superiority; p = 0.3577, ANCOVA; LS Means = -0.377, 95% CI 2-sided [-1.19 to 0.44], Standard Error of Mean 0.407 — [estimate comment as in outcome 1, analysis 1]

44. Secondary Outcome: Changes From Baseline in Visual Analog Scale of Non-Neurological Symptoms. - Dyspnea During Activity (ANCOVA Model)
Description: Clinically significant changes in Visual Analog Scale - Dyspnea during activity. Score ranges from 0 points (no dyspnea) to 10 points (maximum amount of dyspnea)
Time Frame: Baseline (Infusion 1) to Weeks 26 (End of Study)
Measure: Mean (Standard Error); unit: score on a scale (10 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
score on a scale (10 points total) | -1.472 (0.379) | -1.269 (0.405)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; The null hypothesis is that the difference in change from baseline to Weeks 26 in Visual Analog Scale of Non-Neurological Symptoms. - Dyspnea during activity scale score between treatment groups (HB-adMSCs - Placebo) is equal to zero; Test type: Superiority; p = 0.7196, ANCOVA; LS Means = -0.203, 95% CI 2-sided [-1.33 to 0.92], Standard Error of Mean 0.563 — [estimate comment as in outcome 1, analysis 1]

45. Secondary Outcome: Changes From Baseline in Visual Analog Scale of Non-Neurological Symptoms. - Cough (ANCOVA Model)
Description: Clinically significant changes in Visual Analog Scale - Cough. Score ranges from 0 points (no cough) to 10 points (maximum amount of cough).
Time Frame: Baseline (Infusion 1) to Weeks 26 (End of Study)
Measure: Mean (Standard Error); unit: score on a scale (10 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
score on a scale (10 points total) | -0.553 (0.292) | -0.248 (0.312)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; The null hypothesis is that the difference in change from baseline to Weeks 26 in Visual Analog Scale of Non-Neurological Symptoms. - Cough scale score between treatment groups (HB-adMSCs - Placebo) is equal to zero; Test type: Superiority; p = 0.4847, ANCOVA; LS Means = -0.306, 95% CI 2-sided [-1.18 to 0.56], Standard Error of Mean 0.435 — [estimate comment as in outcome 1, analysis 1]

46. Secondary Outcome: Changes From Baseline in Visual Analog Scale of Non-Neurological Symptoms. - Body Aches (ANCOVA Model)
Description: Clinically significant changes in Visual Analog Scale - Body aches. Score ranges from 0 points (no body aches) to 10 points (maximum amount of body aches).
Time Frame: Baseline (Infusion 1) to Weeks 26 (End of Study)
Measure: Mean (Standard Error); unit: score on a scale (10 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
score on a scale (10 points total) | -0.893 (0.446) | -1.511 (0.476)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; The null hypothesis is that the difference in change from baseline to Weeks 26 in Visual Analog Scale of Non-Neurological Symptoms. - Body aches scale score between treatment groups (HB-adMSCs - Placebo) is equal to zero; Test type: Superiority; p = 0.3535, ANCOVA; LS Means = 0.619, 95% CI 2-sided [-0.71 to 1.94], Standard Error of Mean 0.661 — [estimate comment as in outcome 1, analysis 1]

47. Secondary Outcome: Changes From Baseline in Visual Analog Scale of Non-Neurological Symptoms. - Joint Pain (ANCOVA Model)
Description: Clinically significant changes in Visual Analog Scale - Joint Pain. Score ranges from 0 points (no pain) to 10 points (maximum amount of pain).
Time Frame: Baseline (Infusion 1) to Weeks 26 (End of Study)
Measure: Mean (Standard Error); unit: score on a scale (10 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
score on a scale (10 points total) | -1.319 (0.440) | -1.790 (0.470)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; The null hypothesis is that the difference in change from baseline to Weeks 26 in Visual Analog Scale of Non-Neurological Symptoms. - Joint Pain scale score between treatment groups (HB-adMSCs - Placebo) is equal to zero; Test type: Superiority; p = 0.4746, ANCOVA; LS Means = 0.472, 95% CI 2-sided [-0.84 to 1.78], Standard Error of Mean 0.655 — [estimate comment as in outcome 1, analysis 1]

48. Secondary Outcome: Changes From Baseline in Subject's Energy - Fatigue Assessment Form (ANCOVA Model)
Description: Clinically significant changes in Fatigue Assessment form. Total scores can range from 10, indicating the lowest level of fatigue, to 50, denoting the highest.
Time Frame: Baseline (Infusion 1) to Weeks 26 (End of Study)
Measure: Mean (Standard Error); unit: score on a scale (50 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
score on a scale (50 points total) | -8.094 (1.442) | -6.660 (1.538)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; The null hypothesis is that the difference in change from baseline to Weeks 26 in Subject's energy - Fatigue Assessment form scale score between treatment groups (HB-adMSCs - Placebo) is equal to zero; Test type: Superiority; p = 0.5059, ANCOVA; LS Means = -1.433, 95% CI 2-sided [-5.72 to 2.85], Standard Error of Mean 2.141 — [estimate comment as in outcome 1, analysis 1]

49. Secondary Outcome: Changes in Subject's Quality of Life - Short Form 36 Health Survey Questionnaire (General Health)
Description: Short-form (36) Health Survey domain Average General Health; scored on a scale of 0-100; lower score equals more disability.
Time Frame: Baseline (Infusion 1) to Weeks 26 (End of Study)
Measure: Mean (Standard Error); unit: score on a scale (100 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
score on a scale (100 points total) | 6.205 (3.292) | 12.301 (3.520)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; The null hypothesis is that the difference in change from baseline to Weeks 26 in Short Form 36 Health Survey Questionnaire (General Health) between treatment groups (HB-adMSCs - Placebo) is equal to zero; Test type: Superiority; p = 0.2269, ANCOVA; LS Means = -6.095, 95% CI 2-sided [-16.08 to 3.89], Standard Error of Mean 4.990 — [estimate comment as in outcome 1, analysis 1]

50. Secondary Outcome: Changes in Subject's Level of Depression - PHQ 9 Scale.
Description: Clinically significant changes in PHQ (Patient health questionnaire) 9 scale. The PHQ-9 is a 9 question assessment with a total score ranges from 0 to 27 (scores of 5-9 are classified as mild depression; 10-14 as moderate depression; 15-19 as moderately severe depression; ≥ 20 as severe depression) [30].
Time Frame: Baseline (Infusion 1) to Weeks 26 (End of Study)
Measure: Mean (Standard Error); unit: score on a scale (27 points total)
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 39 | 40
score on a scale (27 points total) | -3.666 (0.938) | -3.545 (1.001)
Statistical Analysis 1: Comparison: Treatment vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.8735, ANCOVA; LS Means = -0.122, 95% CI 2-sided [-2.91 to 2.66], Standard Error of Mean 1.392 — [estimate comment as in outcome 1, analysis 1]

51. Secondary Outcome: Changes in Subject's Quality of Life - Short Form 36 Health Survey Questionnaire (Physical Functional Score)
Description: Short-form (36) Health Survey domain Average Physical Functioning; scored on a scale of 0-100; lower score equals more disability.
Time Frame: Baseline (Infusion 1) to Weeks 26 (End of Study)
Measure: Mean (Standard Error); unit: score on a scale (100 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 39 | 40
score on a scale (100 points total) | 13.785 (3.244) | 17.210 (3.461)
Statistical Analysis 1: Comparison: HB-adMSCs vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.4802, ANCOVA; LS Means = -3.424, 95% CI 2-sided [-13.07 to 6.22], Standard Error of Mean 4.820 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Week 0 (Infusion 1) through Week 26 (End of Study)
Arm/Group | HB-adMSCs | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/40
Other Adverse Events (participants affected / at risk) | 34/39 | 28/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HB-adMSCs (N=39) | Placebo (N=40)
Fatigue (General disorders) | 16 (20) | 8 (14)
Influenza like illness (General disorders) | 12 (24) | 4 (6)
Chills (General disorders) | 4 (4) | 0 (0)
Pain (General disorders) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 3 (4) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 16 (25) | 10 (16)
Dizziness (Nervous system disorders) | 3 (4) | 1 (1)
Brain Fog (Nervous system disorders) | 2 (2) | 0 (0)
Cognitive Disorder (Nervous system disorders) | 0 (0) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (2) | 1 (1)
Migraine (Nervous system disorders) | 2 (3) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0)
Anosmia (Nervous system disorders) | 1 (1) | 0 (0)
Coordination abnormal (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Multiple Sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Muscle contractions involuntarily (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 3 (3)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Genital herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Genital infection male (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Post-acute COVID-19 syndrome (Infections and infestations) | 0 (0) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5) | 8 (12)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Infections and infestations) | 1 (1) | 0 (0)
Dyspepsia (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal disorder (Infections and infestations) | 0 (0) | 1 (1)
Paraesthesia oral (Infections and infestations) | 1 (1) | 0 (0)
Toothache (Infections and infestations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Artificial crown procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip surgery (Surgical and medical procedures) | 0 (0) | 1 (2)
Mole excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Oral surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Tongue tie operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Rheumatoid factor positive (Investigations) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sensitive skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eye movement disorder (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT05126563/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT05126563/SAP_001.pdf